CLINICAL TRIAL: NCT02212795
Title: Phase I Study of Pharmacokinetics and Bacteriocidal Activity
Brief Title: Evaluation of Pharmacokinetics Profiles and Bactericidal Activity of Zabofloxacin
Acronym: Bacteriocide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: DW224-I-7
Record Dates: First submitted 2014-07-11; First posted 2014-08-08 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: healthy
MeSH Terms: interventions — zabofloxacin; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A Group (Experimental): 1st oral administration of Zabofloxacin 183mg, 2nd oral administration of Zabofloxacin 367mg and 3rd oral administration of Levofloxacin 250mg
  Interventions: Drug: Zabofloxacin 183mg; Drug: Levofloxacin 250mg; Drug: Zabofloxacin 367mg
- B Group (Experimental): 1st oral administration of Zabofloxacin 367mg, 2nd oral administration of Levofloxacin 250mg and 3rd oral administration of Zabofloxacin 367mg
  Interventions: Drug: Zabofloxacin 183mg; Drug: Levofloxacin 250mg; Drug: Zabofloxacin 367mg
- C Group (Experimental): 1st oral administration of Levofloxacin 250mg, 2nd oral administration of Zabofloxacin 183mg and 3rd oral administration of Zabofloxacin 367mg
  Interventions: Drug: Zabofloxacin 183mg; Drug: Levofloxacin 250mg; Drug: Zabofloxacin 367mg

INTERVENTIONS:
Drug: Zabofloxacin 183mg — Zabofloxacin 183mg single dose
  Other Names: Zabolante 183mg
Drug: Levofloxacin 250mg — Levofloxacin 250mg single dose
  Other Names: Cravit
Drug: Zabofloxacin 367mg — Zabofloxacin 367mg single dose
  Other Names: Zabolante 367mg

SUMMARY:
Phase I clinical study to compare the pharmacokinetic profiles and bactericidal activity of Zabofloxacin 183mg, 367mg and Levofloxacin 250mg after oral administration in healthy volunteer

DETAILED DESCRIPTION:
A Randomized, open label, single dose, crossover phase I clinical study to compare the pharmacokinetic profiles and bactericidal activity of Zabofloxacin 183mg, 367mg and Levofloxacin 250mg after oral administration in healthy volunteer

ELIGIBILITY:
Inclusion Criteria:

* A healthy adult within the range of 19 to 65 years old at the time of screening
* Body Mass Index(BMI)=17.5~30.5kg/m2, one with weight of more than 55kg (BMI= kg/(m)2)
* Congenital or chronic diseases within the last three years, there is no medical examination results of popular characters with no psychotic symptoms or findings
* Doctor checks conducted hematology, blood chemistry, urinalysis and laboratory tests, including an electrocardiogram(EKG) performed during screening tests such as a suitable test subjects who judged
* The purpose of the test participants prior to testing, information, and to hear about the free will fully explain to participate in this study, according to the Institutional Review Board(IRB)-approved consent form signed by the parties in writing

Exclusion Criteria:

* One with clinically significant blood, kidneys, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurological or allergic disease (but ,except for untreated seasonal allergies of asymptomatic at the time of administration) with medical history or evidence
* One with gastrointestinal disease(Such as esophageal stricture or achalasia of the esophagus disease, Crohn disease) to affect drug absorption or surgery(but, excluding simple appendectomy or hernia surgery) with medical history
* Alanine Aminotransferase(ALT) or Aspartate Aminotransferase(AST) > 2 times the upper limit of the normal range
* Within 6 months, 210 g / week of alcohol in excess of a history of regular characters (beer (5%) 1 cup (250 mL) = 10 g, soju(20%) 1 cup (50 mL) = 8 g, Wine (12%) 1 cup (125 mL) = 12 g)
* Take part in other clinical trials within two months
* Systolic Blood Pressure(SBP) ≥ 140 mmHg or Diastolic Blood Pressure (DBP) ≥ 90 mmHg
* The great history of alcohol or drug abuse within 1 year
* Taking medication of drug-metabolizing enzymes that are known to significantly induce or inhibit within 30 days
* More than 20 cigarettes a day smoker
* Taking medication of a prescription drug or nonprescription within 10 days,
* Within two months the whole blood donation have, within one month of the apheresis donation have
* Participate in clinical trials to test drug administration and may be at increased risk due to interpretation of test results, or may interfere with severe supply / chronic medical or mental condition or abnormal laboratory test values in character
* Pregnant women and lactating mothers
* Described lifestyle in this protocol can comply with or can not
* One with other investigator judge to unsuitable

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Cmax and AUC | Predose(0), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 hours
  Maximum of Concentration(Cmax) Area Under Plasma Concentration-Time Curve(AUC)

SECONDARY OUTCOMES:
Pharmacokinetic Profile of Plasma | Predose(0), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 hours
  Maximum drug concentration time(Tmax) Half-time(t1/2) Apparent renal clearance(CL/F) Apparent volume of distribution(Vz/F) Mean of Retention Time(MRT)
Pharmacokinetic Profile of Urine | Predose(-12-0), 0-6, 6-12, 12-24, 24-36, 48-72, 72-96, 96-120 hours
  Umax, Cumulative Amount Excreted(Ae), Fraction of the dose excreted unchanged(fe), Renal Clearance(CLr), Urinary Hydrogen exponent(Urinary pH)
Bactericidal Activity Profile of Urine | Predose(-12-0), 0-6, 6-12, 12-24, 24-36, 48-72, 72-96, 96-120 hours
  Urinary Bactericidal Titers(UBT) Area under the UBT-versus-time curve(AUBT)

CONTACTS AND LOCATIONS:
Overall Officials: MinGul Kim, M.D, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea